CLINICAL TRIAL: NCT06732271
Title: LC-Smart: A Deep Learning-Based Quality Control Model for Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2024-1015-01
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Cholecystectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: Critical view of safety (CVS) is a successful technique to reduce bile duct injury during laparoscopic cholecystectomy (LC). We aimed to create a deep learning-based quality control model for LC and reduce the learning curve for junior surgeons, which would automatically assess whether surgeons are CVS conscious during procedures.Methods: We retrospectively collected 308 LC videos from public datasets (Cholec80, Endoscapes) and Sun Yat-sen Memorial Hospital. Video frames were labeled using binary classification and feature optimization methods, such as black border clipping and sliding windows. Two neural networks, ResNet-50 and EfficientNetV2-S, were trained and evaluated based on F1 scores and accuracy. Additionally, We created an online CVS recognition system (LC-Smart), tested it using 171 films from two hospitals, and compared the results to two local senior doctors.

ELIGIBILITY:
Inclusion Criteria:

* complete video data with no missing footage;
* surgical procedure identified as laparoscopic cholecystectomy;
* full visibility of the surgical area in the video;
* successful completion of the procedure;
* absence of significant anatomical variations
* video resolution no less than 720×560.

Exclusion Criteria:

* substantial intraoperative adhesions
* a history of previous abdominal or pelvic procedures
* a conversion to open surgery during the procedure
* significant bleeding that obscured structural identification.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: people with laparoscopic cholecystectomy
Sampling Method: Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
the surgical time | Nov/2023-Nov/2024

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital,SUn Yat-sen UNiversity, Guangzhou, Guangdong, China